CLINICAL TRIAL: NCT01320449
Title: Identification of New Serum Markers for Detection of Abuse With Erythropoietin
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Aarhus (Other)
Responsible Party: Principal Investigator, Birgitte Nellemann, MD PhDstudent, University of Aarhus
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: M-20110035
Record Dates: First submitted 2011-03-18; First posted 2011-03-22 (Estimated); Last update posted 2012-08-01 (Estimated); Status verified 2012-07

CONDITIONS: Substance Abuse Problem
Keywords: EPO; Proteomics; Carbohydrate metabolism; Fat metabolism; Protein metabolism
MeSH Terms: conditions — Substance-Related Disorders

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (4):
- No training + placebo (Placebo Comparator): 10 young men being investigated with 10 weeks apart. The will receive placebo injections twice a week. Blood samples, blood pressures as well as VO2-max tests will be obtained during the 10 weeks.
  Interventions: Other: Placebo
- No training + EPO (Active Comparator): 10 young men being investigated with 10 weeks apart. During the 10 weeks participants will receive EPO injections twice a week. Blood samples, blood pressures as well as VO2-mas tests will be obtained during the 10 weeks.
  Interventions: Drug: recombinant human erythropoietin
- Training + placebo (Active Comparator): 10 young men will be trained for 10 weeks and investigated before and after. They will receive placebo injections twice a week. Blood samples, blood pressures as well as VO2-max tests will be obtained during the 10 weeks.
  Interventions: Behavioral: Training; Other: Placebo
- Training + EPO (Active Comparator): 10 young men will be investigated with 10 weeks apart. During the ten weeks they will train 3 times a week and receive EPO injections twice a week. Blood samples, blood pressures as well as VO2-max tests will be obtained during the 10 weeks.
  Interventions: Drug: recombinant human erythropoietin; Behavioral: Training

INTERVENTIONS:
Drug: recombinant human erythropoietin — rHuEpo (5000 IU)is administered using a small syringe under the skin every other day for the first 2 weeks, on 3 consecutive days during week 3, and once a week from week 4-10.
  Arms: No training + EPO; Training + EPO
Behavioral: Training — For ten weeks participants will receive supervised endurance training on a bike three times a week. Physical effect will be examined with VO2-max tests before during and after the training period.
  Arms: Training + EPO; Training + placebo
Other: Placebo — placebo (saline) is administered using a small syringe under the skin every other day for the first 2 weeks, on 3 consecutive days during week 3, and once a week from week 4-12.
  Arms: No training + placebo; Training + placebo

SUMMARY:
Epo increases red blood cell production and hence the amount of oxygen that can be transported around the body. It is shown that prolonged use of synthetic Epo (rHuEpo) leads to an increase in the period of time a given physical work can be performed, therefore it will continue to be abused by athletes, especially in endurance sports.

The existing method for measuring the abuse of rHuEpo approved by the World Anti-Doping Agency (WADA) is based on differences in the sugar groups bound to rHuEpo and Epo produced in the body, respectively.

Proteomics is a method by which one can look at all the proteins in blood at the same time. Even proteins that have changed very little can be distinguished. The main objective of this project is to investigate the effect of prolonged treatment with rHuEpo on changes in blood proteins in healthy young men.

ELIGIBILITY:
Inclusion Criteria:

* healthy men
* age 18-35
* untrained
* BMI: 20-25

Exclusion Criteria:

* smokers
* chronic diseases
* malignancy (former or present)
* alcohol, drug or EPO abuse

Ages: 18 Years to 35 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 35 (Actual)
Dates: Start 2011-08; Primary Completion 2012-07 (Actual); Study Completion 2012-07 (Actual)

PRIMARY OUTCOMES:
Changes in serum protein isoforms measured by proteomics | 10 months
  We wish to identify proteins or isoforms hereof that change with rHuEpo treatment, in order to identify new biomarkers in the blood that can be used to detect rHuEpo abuse.

SECONDARY OUTCOMES:
Changes in substrate metabolism in relation to rHuEpo treatment and endurance training | 10 months
  Metabolic and mechanistic effects of 10 weeks of training and use of EPO on fat and skeletal muscle tissue as well as on a whole body level. A variety of different tracers and indirect calorimetry will be used.

CONTACTS AND LOCATIONS:
Overall Officials: Britt Christensen, M.Sc., PhD, Principal Investigator — Aarhus University Hospital
Locations (2):
- Denmark (2):
  - Aarhus University Hospital, Aarhus, Aarhus
  - Department of Endocrinology, Research Laboratories, Aarhus

REFERENCES:
- [Derived] Larsen MS, Holm L, Svart MV, Hjelholt AJ, Bengtsen MB, Dollerup OL, Dalgaard LB, Vendelbo MH, van Hall G, Moller N, Mikkelsen UR, Hansen M. Effects of protein intake prior to carbohydrate-restricted endurance exercise: a randomized crossover trial. J Int Soc Sports Nutr. 2020 Jan 28;17(1):7. doi: 10.1186/s12970-020-0338-z. PMID 31992300
- [Derived] Nielsen J, Christensen AE, Nellemann B, Christensen B. Lipid droplet size and location in human skeletal muscle fibers are associated with insulin sensitivity. Am J Physiol Endocrinol Metab. 2017 Dec 1;313(6):E721-E730. doi: 10.1152/ajpendo.00062.2017. Epub 2017 Jul 25. PMID 28743757
- [Derived] Christensen B, Ludvigsen M, Nellemann B, Kopchick JJ, Honore B, Jorgensen JO. Serum proteomic changes after randomized prolonged erythropoietin treatment and/or endurance training: detection of novel biomarkers. PLoS One. 2015 Feb 13;10(2):e0117119. doi: 10.1371/journal.pone.0117119. eCollection 2015. PMID 25679398